CLINICAL TRIAL: NCT01325168
Title: The Effect of Intranasal Oxytocin on Emphatic Abilities in Patients With PTSD
Brief Title: The Effect of Intranasal Oxytocin on Emphatic Abilities in Patients With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0085-11CTIL
Record Dates: First submitted 2011-03-20; First posted 2011-03-29 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; empathy; oxytocin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): 32 PTSD patients intervention: Drug: syntocinon nasal spray / placebo nasal spray nasal OT - 24 IU, 3 inhalations of 4IU to each nostril (45 sec waiting between the inhalations)
  Interventions: Drug: syntocinon nasal spray; Drug: placebo nasal spray
- control group (Other): control group - 30 healthy control subjects intervention: Drug: syntocinon nasal spray / placebo nasal spray nasal OT - 24 IU, 3 inhalations of 4IU to each nostril (45 sec waiting between the inhalations)
  Interventions: Drug: syntocinon nasal spray; Drug: placebo nasal spray

INTERVENTIONS:
Drug: syntocinon nasal spray — nasal oxytocin - 24 IU, 3 inhalations of 4IU to each nostril (45 sec waiting between the inhalations)
  Other Names: nasal oxytocin - 24 IU,
Drug: placebo nasal spray — nasal placebo - 24 IU, 3 inhalations of 4IU to each nostril (45 sec waiting between the inhalations)
  Other Names: nasal placebo - 24 IU,

SUMMARY:
Oxytocin (OT) - a neurohormone and neuromodulator which is mainly synthesized in the hypothalamus - is a key mediator of complex social and affective behaviors, including emotional empathy. Recently, several theoretical studies suggested that PTSD patients have abnormal functioning of the OT system. According to these theories, dysfunction in the oxytocin system may modulate the interpersonal impairment that characterizes PTSD, and therefore intranasal OT may potentially relieve these symptoms. The main goal of this study is to examine the effects of administration of nasal OT on empathic abilities among PTSD patients. Another goal of this study is to examine the relationship between empathic abilities and the ability to retrieve autobiographical memories among PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

* PTSD patients (DSM-IV criteria)
* Ability to provide written informed consent

Exclusion Criteria:

* Suicidality
* Psychosis
* Arrhythmia
* Cardiac disease (arrythmia, heart failure)
* Hyponatremia
* Severe renal insufficiency
* Liver cirrhosis
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Computer tasks that assess empathy, Another goal of this study is to examine the relationship between empathic abilities and the ability to retrieve autobiographical memories among PTSD patients. | 1 hour after the inhalation the OT
  The computer tasks will assess emotional empathy(e.g. task that assess the ability to recognizes emotional facial expressions ('face morphing'), and task that assess the ability to recognizes emotions depicted in a biological motion ('biological motion')), And cognitive empathy ( task that assess the ability to judge mental states based on verbal and eye gaze cues (ToM task)).

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, MD., Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam health care campus, Haifa
  - Rambam Medical Center, Haifa